CLINICAL TRIAL: NCT05927675
Title: Dynamic Profiling of Microbiome and Metabolites Regarding Physical Activity in Middle-aged Korean Women
Brief Title: Changes in Microbiome and Metabolites Regarding Physical Activity in Middle-aged Korean Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University (Other)
Responsible Party: Principal Investigator, JiYeob Choi, Professor, Seoul National University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PA-1812-129-997
Record Dates: First submitted 2023-06-13; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Healthy
Keywords: Microbiome; Metabolite; Physical activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise intervention (Experimental)
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — The exercise intervention program consisted of two distinct periods. During period 1, subjects participated in a moderate to vigorous intensity exercise program for 40 minutes a day, 4 days a week. The exercise program was conducted in Tabata format targeting 70% of the maximum heart rate. Recovery was then induced for 1 minute and 30 seconds, allowing the heart rate to return to resting levels. The exercise routine primarily consisted of full-body exercises, functional training, and power exercises.
  During period 2, a low-intensity static exercise program was implemented. Similar to period 1, the subjects exercised for 40 minutes a day, 4 days a week. The exercise program included static exercises. The maximum heart rate was maintained below 50%. The detailed exercise program consisted of stretching movements and balance movements.

SUMMARY:
This study aimed to examine the effect of physical activity (PA) on health through changes in multi-omics biomarkers during 6 months of exercise intervention.

DETAILED DESCRIPTION:
This study aimed to examine the effect of physical activity (PA) on health through changes in multi-omics biomarkers during 6 months of exercise intervention. Twenty-seven healthy middle-aged women were recruited and 14 subjects completed the exercise intervention. A total of three blood and stool samples were collected at 3-month intervals. The amount of PA was measured with an accelerometer. Clinical variables were used, including blood pressure, grip strength, flexibility, and blood glucose levels and lipid markers obtained from laboratory tests. The concentration of blood metabolites was measured by targeted metabolomics. Fecal microbiome data were obtained by 16S rRNA gene amplicon sequencing. During the second half period (period 2), Coronavirus disease 2019 (COVID-19) occurred and spread out in Korea, and PA decreased compared with the first half period (period 1). Blood pressure, hemoglobin A1c (HbA1c), and low-density lipoprotein cholesterol (LDL-C) decreased in period 1 and tended to increase again during period 2. Forty metabolites were changed significantly during period 1, and investigators found that 6 of them were correlated with changes in blood pressure, HbA1c, and LDL-C via network analysis. Our results may suggest the relationship between changes in biomarkers at multi-omics levels during exercise and a message that reduced PA due to COVID-19 can adversely affect health.

ELIGIBILITY:
Inclusion Criteria:

* age 40 - 59 (middled aged women)
* Those who have no difficulties in daily living
* Those who engage in sedentary activities most of the day
* Willing to commit throughout the study

Exclusion Criteria:

* Antibiotics medication in the last month.
* Those who are in the treatment of the following diseases: Liver disease, Neurological disease, Respiratory disease, Tumors, Psychiatric disorders, Angina, Myocardial infarction, and Stroke

Ages: 40 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
Change in Systolic blood pressure (SBP) between baseline and 3rd month | baseline ~ 3 month
  blood pressure (mmHg) (Omron Corporation, Kyoto, Japan)
Change in Systolic blood pressure (SBP) between 3rd month and 6th month | 3 ~ 6 month
  blood pressure (mmHg) (Omron Corporation, Kyoto, Japan)
Changes in diastolic blood pressure (DBP) between baseline and 3rd month | baseline ~ 3 month
  blood pressure (mmHg) (Omron Corporation, Kyoto, Japan)
Changes in diastolic blood pressure (DBP) between 3rd month and 6th month | 3 ~ 6 month
  blood pressure (mmHg) (Omron Corporation, Kyoto, Japan)
Changes in hemoglobin A1c (HbA1c) between baseline and 3rd month | baseline ~ 3 month
  The concentrations of hemoglobin A1c (HbA1c) (mg/dL) (HLC-723G11 analyzer, TOSOH kabushiki kaisha, HPLC)
Changes in hemoglobin A1c (HbA1c) between 3rd month and 6th month | 3 ~ 6 month
  The concentrations of hemoglobin A1c (HbA1c) (mg/dL) (HLC-723G11 analyzer, TOSOH kabushiki kaisha, HPLC)
Changes in total cholesterol between baseline and 3rd month | baseline ~ 3 month
  total cholesterol (mg/dL) (Cobas C701/702 autochemistry analyzer, Roche, enzyme method)
Changes in total cholesterol between 3rd month and 6th month | 3 ~ 6 month
  total cholesterol (mg/dL) (Cobas C701/702 autochemistry analyzer, Roche, enzyme method)
Changes in high-density lipoprotein cholesterol (HDL-C) between baseline and 3rd month | baseline ~ 3 month
  high-density lipoprotein cholesterol (HDL-C) (mg/dL) (Cobas C701/702 autochemistry analyzer, Roche, enzyme method)
Changes in high-density lipoprotein cholesterol (HDL-C) between 3rd month and 6th month | 3 ~ 6 month
  high-density lipoprotein cholesterol (HDL-C) (mg/dL) (Cobas C701/702 autochemistry analyzer, Roche, enzyme method)
Changes in low-density lipoprotein cholesterol (LDL-C) betweenbaseline and 3rd month | baseline ~ 3 month
  low-density lipoprotein cholesterol (LDL-C) (mg/dL) (Cobas C701/702 autochemistry analyzer, Roche, enzyme method)
Changes in low-density lipoprotein cholesterol (LDL-C) between 3rd month and 6th month | 3 ~ 6 month
  low-density lipoprotein cholesterol (LDL-C) (mg/dL) (Cobas C701/702 autochemistry analyzer, Roche, enzyme method)
Changes in Microbiome between baseline and 3rd month | baseline ~ 3 month
  The composition of the gut microbiome obtained by 16S rRNA gene amplicon sequencing.
Changes in Microbiome between 3rd month and 6th month | 3 ~ 6 month
  The composition of the gut microbiome obtained by 16S rRNA gene amplicon sequencing.
Changes in Metabolome between baseline and 3rd month | baseline ~ 3 month
  Plasma metabolite concentrations were measured by using the AbsoluteIDQ p 180 kit and the Bile acids kit.
Changes in Metabolome between 3rd month and 6th month | 3 ~ 6 month
  Plasma metabolite concentrations were measured by using the AbsoluteIDQ p 180 kit and the Bile acids kit.

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Yeob Choi, Principal Investigator — Seoul National University
Locations (1):
- Seoul National University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park J, Kim J, Kang J, Choi J, Kim JE, Min KJ, Choi SW, Cho JY, Lee M, Choi JY. A 6-month exercise intervention clinical trial in women: effects of physical activity on multi-omics biomarkers and health during the first wave of COVID-19 in Korea. BMC Sports Sci Med Rehabil. 2024 Jan 29;16(1):30. doi: 10.1186/s13102-024-00824-6. PMID 38287431